CLINICAL TRIAL: NCT00034255
Title: Single Dose and 34-Day Tolerance Study of INGAP Peptide in Insulin Deficient Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GMP Endotherapeutics (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: INGAP-01-001
Record Dates: First submitted 2002-04-24; First posted 2002-04-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-06

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — INGAP peptide

INTERVENTIONS:
Drug: INGAP Peptide

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single and multiple doses of intramuscular INGAP Peptide given for the first time in humans as a potential treatment for diabetes.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting all of the following inclusion criteria at screening can be considered for admission to the study.

Stage 1 and Stage 2:

1. Male and female patients with, type 1 diabetes mellitus that are 18 through 70 years of age, or type 2 diabetes mellitus that are 30 through 70 years of age.
2. Patients who are insulin deficient and are diagnosed with type 1 or type 2 diabetes mellitus, and are currently well managed with insulin, with or without metformin.
3. Patients who have been on stable doses of insulin treatment for 90 days prior to study randomization.

Exclusion Criteria:

Patients meeting any of the following exclusion criteria at screening will not be enrolled in the study:

1. Patients with a history of any clinically significant retinopathy, symptomatic autonomic neuropathy, unstable angina, or kidney problems.
2. Patients with an uncontrolled or untreated significant pulmonary, neurological condition, or cardiovascular disease, including hypertension, congestive heart failure, angina, or peripheral vascular disease.
3. Patients who have received any investigational product within 30 days of admission into the study.
4. Patients with a history or clinical evidence of multiple organ autoimmune disorders.
5. Patients with a medical condition, serious intercurrent illness, or extenuating circumstance that would significantly decrease study compliance, including all prescribed follow-up.
6. Patients who are lactating and breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62
Dates: Start 2001-12

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - VASDHS Medical Center, San Diego, California
  - MedStar Research Institute - Clinical Research Center, Washington D.C., District of Columbia
  - UNC Diabetes, Endocrinology, Metabolism Clinic, Durham, North Carolina
  - Texas Diabetes Institute, San Antonio, Texas